CLINICAL TRIAL: NCT05320341
Title: The Effects of Total Intravenous and Inhalation Anesthesia Maintenance on Tissue Oxygenation in Coronary Artery Bypass Graft Surgery
Brief Title: TIVA Versus Inhalational Anesthesia and Tissue Oxygenation in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Eda Balci, Medical Doctor, Ankara City Hospital Bilkent
Other Study IDs: MH.2.5
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Cardiac Anesthesia
Keywords: tissue oxygenation; total intravenous anesthesia; inhalational anesthesia; cardiac surgery; NIRS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TIVA group: During the anesthesia maintenance of the TIVA group, 3 μg.kg-1 fentanyl, 0.01-0.05 mg.kg-1 midazolam, and 0.2 mg.kg-1 rocuronium bromide were applied throughout the operation to keep BIS between 40 and 60, approximately once every 45 minutes.
  Interventions: Procedure: TIVA
- SEVO group: During the anesthesia maintenance of the SEVO group, 2-3% sevoflurane (1-2 MAC), 3 μg.kg-1 fentanyl and 0.2 mg.kg-1 rocuronium bromide were applied throughout the operation to keep BIS between 40-60.
  Interventions: Procedure: SEVO

INTERVENTIONS:
Procedure: TIVA — During the anesthesia maintenance of the TIVA group, 3 μg.kg-1 fentanyl, 0.01-0.05 mg.kg-1 midazolam, and 0.2 mg.kg-1 rocuronium bromide were applied throughout the operation to keep BIS between 40 and 60, approximately once every 45 minutes.
  Groups: TIVA group
Procedure: SEVO — During the anesthesia maintenance of the SEVO group, 2-3% sevoflurane (1-2 MAC), 3 μg.kg-1 fentanyl and 0.2 mg.kg-1 rocuronium bromide were applied throughout the operation to keep BIS between 40-60.
  Groups: SEVO group

SUMMARY:
The aim of this study was to evaluate the effect of total intravenous anesthesia (TIVA) and inhalational anesthesia techniques on tissue oxygenation in cardiac surgery. The primary objective of this study was to compare the effects of midazolam-based TIVA and sevoflurane-based (SEVO) inhalation anesthesia maintenance on intraoperative central and regional tissue oxygenation parameters.

DETAILED DESCRIPTION:
A pressing issue in anesthesiology involves developing an understanding of the non-anesthetic effects of the medications typically used in intravenous and inhalation anesthesia methods. Few studies describe the effects of both intravenous and inhalational anesthetics on regional tissue perfusion is described under stable anesthetic conditions. There is the issue of whether inhalational anesthetics compromise regional tissue perfusion even though systemic parameters are within normal ranges. It is still debated how these effects may be different under pathophysiological conditions, such as cardiac surgery.

Maintaining tissue perfusion and oxygenation is the cornerstone of therapy for patients with cardiac disease. An imbalance in oxygen delivery and tissue oxygen consumption leads to anaerobic metabolism, cellular injury, and organ dysfunction, and is associated with poor outcomes. Consequently, monitoring tissue oxygen delivery and consumption status is of paramount importance in cardiac surgery patients. Routinely used monitors in intraoperative settings such as pulse oximetry, blood pressures, hemoglobin saturation levels, lactate, acid-base status, and central venous oxygen saturation levels all reflect tissue metabolism. Near-infrared spectroscopy (NIRS) is a non-invasive optical technique that can be used to continuously monitor tissue oxygen delivery and oxygen consumption status. Cerebral autoregulation can blunt the effect of impaired systemic oxygen delivery. Thus, cerebral NIRS may be a good predictor of neurological outcomes, but skeletal muscle NIRS serves as a follow-up indicator of many other postoperative complications due to impaired perfusion and oxygenation. Therefore, both cerebral and somatic monitoring may contribute to a more complete evaluation of hemodynamic competence. Obtaining the cerebral and somatic oxygenation levels are valuable to help in clinical management during cardiopulmonary bypass (CPB) and cardiac surgery as a whole.

The aim of this study was to evaluate the effect of total intravenous anesthesia (TIVA) and inhalational anesthesia techniques on tissue oxygenation in cardiac surgery. For this purpose, the effects of midazolam-based TIVA or sevoflurane-based inhalation anesthesia maintenance on intraoperative central and somatic tissue oxygenation parameters were compared in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

- coronary surgeries with CPB

Exclusion Criteria:

* emergency surgeries,
* operations
* ejection fraction under 40%
* coronary surgeries in conjunction with other procedures
* cerebrovascular accident
* neurological disorders
* hematologic disorder
* chronic alcohol use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who undergoing coronary surgeries with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Hemodynamic parameters | 5 minutes after anesthesia induction
  mean arterial pressure in mmHg was recorded
Hemodynamic parameters | 5 minutes after anesthesia induction
  heart rate (beat per minute) were recorded
Hemodynamic parameters | After cardiopulmonary bypass cannulation, an average of 5 minutes
  mean arterial pressure (mmHg) was recorded
Hemodynamic parameters | After cardiopulmonary bypass cannulation, an average of 5 minutes
  heart rate (beat per minute) was recorded
Hemodynamic parameters | 10th minute of cardiopulmonary bypass
  mean arterial pressure (mmHg) was recorded
Hemodynamic parameters | 10th minute of cardiopulmonary bypass
  heart rate (beat per minute) was recorded
Hemodynamic parameters | 10 minutes after cross clamp removal
  mean arterial pressure (mmHg) was recorded
Hemodynamic parameters | 10 minutes after cross clamp removal
  heart rate (beat per minute) was recorded
Hemodynamic parameters | 10 minutes after CPB completion
  mean arterial pressure (mmHg) was recorded
Hemodynamic parameters | 10 minutes after CPB completion
  heart rate (beat per minute ) was recorded
Hemodynamic parameters | upon sternum closing
  mean arterial pressure (mmHg) was recorded
Hemodynamic parameters | upon sternum closing
  heart rate (beat per minute) was recorded
Arterial gas sampling | 5 minutes after anesthesia induction
  pH levels were recorded
Arterial gas sampling | 5 minutes after anesthesia induction
  central venous saturation (%) levels were recorded
Arterial gas sampling | 5 minutes after anesthesia induction
  lactate levels (mmol/L) were recorded
Arterial gas sampling | 5 minutes after anesthesia induction
  Hemoglobin (g/dL) levels were recorded
Arterial gas sampling | After cardiopulmonary bypass cannulation, an average of 5 minutes
  pH levels were recorded
Arterial gas sampling | After cardiopulmonary bypass cannulation, an average of 5 minutes
  central venous saturation (%) levels were recorded
Arterial gas sampling | After cardiopulmonary bypass cannulation, an average of 5 minutes
  lactate (mmol/L) levels were recorded
Arterial gas sampling | After cardiopulmonary bypass cannulation, an average of 5 minutes
  hemoglobin (g/dL)levels were recorded
Arterial gas sampling | 10th minute of cardiopulmonary bypass
  pH levels were recorded
Arterial gas sampling | 10th minute of cardiopulmonary bypass
  central venous saturation (%) levels were recorded
Arterial gas sampling | 10th minute of cardiopulmonary bypass
  lactate (mmol/L) levels were recorded
Arterial gas sampling | 10th minute of cardiopulmonary bypass
  hemoglobin (g/dL) levels were recorded
Arterial gas sampling | 10 minutes after cross clamp removal
  pH levels were recorded
Arterial gas sampling | 10 minutes after cross clamp removal
  central venous saturation (%) levels were recorded
Arterial gas sampling | 10 minutes after cross clamp removal
  lactate (mmol/L) levels were recorded
Arterial gas sampling | 10 minutes after cross clamp removal
  hemoglobin (g/dL) levels were recorded
Arterial gas sampling | 10 minutes after CPB completion
  pH levels were recorded
Arterial gas sampling | 10 minutes after CPB completion
  central venous saturation (%) levels were recorded
Arterial gas sampling | 10 minutes after CPB completion
  lactate (mmol/L) levels were recorded
Arterial gas sampling | 10 minutes after CPB completion
  hemoglobin (g/dL) levels were recorded
Arterial gas sampling | upon sternum closing
  pH levels were recorded
Arterial gas sampling | upon sternum closing
  central venous saturation (%) levels were recorded
Arterial gas sampling | upon sternum closing
  lactate (mmol/L) levels were recorded
Arterial gas sampling | upon sternum closing
  hemoglobin (g/dL) levels were recorded
NIRS | 5 minutes after anesthesia induction
  cerebral (rSO2) values were recorded
NIRS | 5 minutes after anesthesia induction
  somatic (rSO2) values were recorded
NIRS | After cardiopulmonary bypass cannulation, an average of 5 minutes
  cerebral (rSO2) values were recorded
NIRS | After cardiopulmonary bypass cannulation, an average of 5 minutes
  somatic(rSO2) values were recorded
NIRS | 10th minute of cardiopulmonary bypass
  cerebral (rSO2) values were recorded
NIRS | 10th minute of cardiopulmonary bypass
  somatic (rSO2) values were recorded
NIRS | 10 minutes after cross clamp removal
  cerebral (rSO2) were recorded
NIRS | 10 minutes after cross clamp removal
  somatic (rSO2) were recorded
NIRS | 10 minutes after CPB completion
  cerebral(rSO2)values were recorded
NIRS | 10 minutes after CPB completion
  somatic (rSO2) values were recorded
NIRS | upon sternum closing
  cerebral(rSO2)values were recorded
NIRS | upon sternum closing
  somatic (rSO2) values were recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Select State/Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Turek Z, Sykora R, Matejovic M, Cerny V. Anesthesia and the microcirculation. Semin Cardiothorac Vasc Anesth. 2009 Dec;13(4):249-58. doi: 10.1177/1089253209353134. Epub 2009 Dec 2. PMID 19959497
- [Result] Bickler P, Feiner J, Rollins M, Meng L. Tissue Oximetry and Clinical Outcomes. Anesth Analg. 2017 Jan;124(1):72-82. doi: 10.1213/ANE.0000000000001348. PMID 27308951
- [Result] De Backer D, Dubois MJ, Schmartz D, Koch M, Ducart A, Barvais L, Vincent JL. Microcirculatory alterations in cardiac surgery: effects of cardiopulmonary bypass and anesthesia. Ann Thorac Surg. 2009 Nov;88(5):1396-403. doi: 10.1016/j.athoracsur.2009.07.002. PMID 19853081